CLINICAL TRIAL: NCT04055558
Title: Lymphoproliferative Disorders After Diagnosis of Childhood Acute Lymphoblastic Leukemia/Lymphoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Collaborators: Israeli Society for Pediatric Hematology-Oncology (Other); International BFM Study Group (Network)
Responsible Party: Sponsor
Other Study IDs: RMC-0109-17
Record Dates: First submitted 2019-08-11; First posted 2019-08-13 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-08

CONDITIONS: Childhood Leukemia and Lymphoma
Keywords: childhood leukemia; lymphoproliferative disorders; EBV
MeSH Terms: conditions — Lymphoma; Lymphoproliferative Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lymphoproliferative disorders (LPD) are a major cause of morbidity and mortality in immunodeficient patients. There have been isolated case reports of patients with childhood ALL who developed LPD after ALL diagnosis, without undergoing stem cell transplantation, but data regarding such cases are limited. We propose here an international collaboration, to form a comprehensive database of children who developed LPD after diagnosis of acute lymphoblastic leukemia/lymphoma

DETAILED DESCRIPTION:
Lymphoproliferative disorders (LPD) are a major cause of morbidity and mortality in immunodeficient patients. These disorders have been extensively described in the post-transplant setting, ie after hematopoietic stem cell (SCT) or solid organ (SOT) transplant. However, since the 1980's, there have been isolated case reports of patients with childhood ALL, who developed LPD after diagnosis of ALL, without undergoing SCT. Comprehensive information is unavailable regarding the prevalence, clinical manifestations, treatment, outcome and pathogenesis of such disorders in this setting. We propose here an international collaboration, to form a comprehensive database of children who developed LPD during the treatment of acute lymphoblastic leukemia/lymphoma (ALL/LBL).

Information will be collected in a de-identified fashion regarding patient characteristics, leukemia and LPD characteristics, treatment and outcome. The aims of this retrospective study are:

1. To build a database of children who developed LPD after diagnosis of ALL/LBL
2. To investigate the characteristics and outcome of this disorder

ELIGIBILITY:
Inclusion Criteria:

* Children and young adults treated for acute lymphoblasticleukemia/lymphoma who developed LPD after ALL/LBL diagnosis

Exclusion Criteria:

* age>30 years

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and young adults (<30 years of age), previously diagnosed with acute lymphoblastic leukemia/lymphoma, who developed LPD after ALL/LBL diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-08-25 (Actual); Primary Completion 2021-12-18 (Estimated); Study Completion 2022-03-18 (Estimated)

PRIMARY OUTCOMES:
Probability of survival | 1 year
  Assess six-month probability of survival since LPD diagnosis

SECONDARY OUTCOMES:
Event-free survival | 5 years
  Assess 5-year event-free survival since acute lymphoblastic leukemia/lymphoma diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Elitzur, MD, Principal Investigator — Schneider Children's Medical Center
Locations (1):
- Schneider Children's Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: Undecided